CLINICAL TRIAL: NCT04205487
Title: PrEP Readiness Interventions for Supporting Motivation in Stimulant-Using Sexual Minority Men
Brief Title: PrEP Readiness Interventions for Supporting Motivation
Acronym: PRISM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: City University of New York (Other); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Carrico, PhD, Professor and Chair, Florida International University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 20180823; R34DA046367 (NIH)
Record Dates: First submitted 2019-12-13; First posted 2019-12-19 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: HIV Infections; Pre-exposure Prophylaxis; Substance Use Disorders
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial (SMART)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Contingency Management (CM) - Only (Non-Responder) (Experimental): Non-responders to CM financial inancial incentives for PrEP clinical evaluation and filling a PrEP prescription in Stage 1 that were randomized to assessments only in Stage 2.
  Interventions: Behavioral: Contingency Management (CM)
- Motivational Interviewing (MI) - Only (Non-Responder) (Experimental): Non-responders to two MI sessions focusing on stimulant use, sexual risk, and PrEP use in Stage 1 that were randomized to assessments only in Stage 2
  Interventions: Behavioral: Motivational Interviewing (MI)
- CM+MI (Experimental): Non-responders CM financial incentives for PrEP clinical evaluation and filling a PrEP prescription in Stage 1 that were randomized to receive two sessions of MI in Stage 2.
  Interventions: Behavioral: Motivational Interviewing (MI); Behavioral: Contingency Management (CM)
- MI+CM (Experimental): Non-responders to two MI sessions focusing on stimulant use, sexual risk, and PrEP use in Stage 1 that were randomized to receive CM financial incentives for PrEP clinical evaluation and filling a PrEP prescription in Stage 2.
  Interventions: Behavioral: Motivational Interviewing (MI); Behavioral: Contingency Management (CM)
- CM-Only (Responder) (Experimental): Respnders to CM financial incentives for CM will include financial incentives for rEP clinical evaluation and filling a PrEP prescription in Stage 1.
  Interventions: Behavioral: Contingency Management (CM)
- MI-Only (Responder) (Experimental): Responders to two MI sessions focusing on stimulant use, sexual risk, and PrEP use will be delivered in Stage 1.
  Interventions: Behavioral: Motivational Interviewing (MI)

INTERVENTIONS:
Behavioral: Motivational Interviewing (MI) — Two motivational interviewing sessions focusing on stimulant use, sexual risk, and PrEP uptake will be delivered via Zoom.
  Arms: CM+MI; MI+CM; MI-Only (Responder); Motivational Interviewing (MI) - Only (Non-Responder)
Behavioral: Contingency Management (CM) — CM will include financial incentives for PrEP clinical evaluation and filling a PrEP prescription.
  Arms: CM+MI; CM-Only (Responder); Contingency Management (CM) - Only (Non-Responder); MI+CM

SUMMARY:
The overarching goal of this formative research is to examine whether, and in what combination, contingency management (CM) and motivational interviewing (MI) can facilitate entry of stimulant-using men who have sex with men (MSM) into the pre-exposure prophylaxis (PrEP) care continuum.

DETAILED DESCRIPTION:
In Stage 1, participants will be randomized to receive either: 1) three months of CM; or 2) two sessions of MI. All participants will be assessed at three months post-randomization for non-response. In Stage 2, a second randomization where non-responders (i.e., those who have not filled a PrEP prescription) are assigned to: 1) Switch to sequentially receive the other intervention (i.e., CM+MI or MI+CM); or 2) Continue with assessments only (i.e., CM-Only or MI-Only). All participants will complete a final assessment at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Sexually active cisgender sexual minority man
* Reports using stimulants in the past three months
* HIV-negative serostatus
* Meets Centers for Disease Control and Prevention (CDC) criteria for PrEP eligibility

Exclusion Criteria:

* Currently prescribed PrEP
* Unable to provide informed consent
* Severe psychiatric symptoms (e.g., mania, psychosis) that impair capacity to participate

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 70 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam W Carrico, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami School of Medicine, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Davis Ewart L, Larson ME, Ghanooni D, Verhagen R, Manuel J, McCollister K, Fardone E, DeVries B, Dilworth S, Blackstock M, Doblecki-Lewis S, Nahum-Shani I, Grov C, Carrico AW. Getting to yes: Pilot sequential multiple assignment randomized trial of motivational enhancement interventions targeting preexposure prophylaxis use in sexual minority men who use stimulants. Health Psychol. 2025 Mar;44(3):310-320. doi: 10.1037/hea0001489. PMID 39992777
- [Derived] Davis-Ewart L, Grov C, Verhagen R, Manuel J, Viamonte M, Dilworth S, O'Dell N, Valentin O, Carr S, Cherenack E, Henderson C, Doblecki-Lewis S, Nahum-Shani I, Carrico AW. Motivational Enhancement Interventions to Increase Pre-Exposure Prophylaxis Use in Sexual Minority Men Who Use Stimulants: Protocol for a Pilot Sequential Multiple Assignment Randomized Trial. JMIR Res Protoc. 2023 Oct 13;12:e48459. doi: 10.2196/48459. PMID 37831485
- [Derived] Davis-Ewart L, Grov C, Verhagen R, Manuel J, Viamonte M, Dilworth S, Valentin O, Cherenack EM, Carr S, Doblecki-Lewis S, Nahum-Shani I, Carrico AW. Randomized Controlled Trial of Motivational Enhancement Interventions to Increase Pre-Exposure Prophylaxis Use in Sexual Minority Men Who Use Stimulants. Res Sq [Preprint]. 2023 Apr 20:rs.3.rs-2787003. doi: 10.21203/rs.3.rs-2787003/v1. PMID 37131755
- [Derived] Davis-Ewart L, Lee JY, Viamonte M, Colon-Burgos J, Harkness A, Kanamori M, Duncan DT, Doblecki-Lewis S, Carrico AW, Grov C. "The familiar taste of poison": a qualitative study of multi-level motivations for stimulant use in sexual minority men living in South Florida. Harm Reduct J. 2023 Apr 26;20(1):58. doi: 10.1186/s12954-023-00787-w. PMID 37101251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A US national sample of sexual minority men taking pre-exposure prophylaxis (PrEP) who reported using stimulants (i.e., methamphetamine, powder cocaine, or crack-cocaine) in the past three months was recruited from social networking applications and existing consent-to-contact databases.
Pre-assignment Details: Participants completed a run-in period where they were asked to provide a saliva sample via mail to confirm they were not living with HIV. Those who did not provide a saliva sample or those with reactive HIV results were excluded.
Groups:
- Contingency Management (CM) - Only (Non-Responder or Lost to Follow Up During Stage 1): Participants randomized in Stage 1 to receive CM financial incentives for PrEP clinical evaluation and filling a PrEP prescription that were non-responders. These participants were randomized to receive assessments only in Stage 2, or were lost to follow up during Stage 1 and we not re-randomized during Stage 2.
- Motivational Interviewing (MI) - Only (Non-Responder or Lost to Follow Up During Stage 1): Participants randomized in Stage 1 two MI sessions focusing on stimulant use, sexual risk, and PrEP uptake delivered via Zoom.. These participants were randomized to receive assessments only in Stage 2, or were lost to follow up during stage 1 and were not re-randomized during Stage 2.
- CM+MI: Sequential delivery of CM(Stage 1) and then MI (Stage 2) for non-responders at the stage-two randomization to "switch."
- MI+CM: Sequential delivery of MI (Stage 1) and then CM (Stage 2) for non-responders at the stage-two randomization to "switch."
- CM-Only (Responder): Responders randomized to receive CM financial incentives for PrEP clincial evaluation and uptake in Stage 1 who provided evidence of a recent PrEP prescription.
- MI-Only (Responder): Responders randomized to receive two MI sessions focusing on stimulant use, sexual risk, and PrEP uptake delivered via Zoom.
Period: First Stage Intervention (Months 1-3)
Arm/Group | Contingency Management (CM) - Only (Non-Responder or Lost to Follow Up During Stage 1) | Motivational Interviewing (MI) - Only (Non-Responder or Lost to Follow Up During Stage 1) | CM+MI | MI+CM | CM-Only (Responder) | MI-Only (Responder)
Started | 15 | 21 | 9 | 7 | 11 | 7
Completed | 5 | 13 | 9 | 7 | 11 | 7
Not Completed | 10 | 8 | 0 | 0 | 0 | 0
Period: Second Stage Intervention (Months 4-6)
Arm/Group | Contingency Management (CM) - Only (Non-Responder or Lost to Follow Up During Stage 1) | Motivational Interviewing (MI) - Only (Non-Responder or Lost to Follow Up During Stage 1) | CM+MI | MI+CM | CM-Only (Responder) | MI-Only (Responder)
Started | 5 | 13 | 9 | 7 | 11 | 7
Completed | 3 | 12 | 9 | 7 | 7 | 7
Not Completed | 2 | 1 | 0 | 0 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- CM-Only (Non-Responder): Participants randomized in Stage 1 to receive CM financial incentives for PrEP clinical evaluation and filling a PrEP prescription that were non-responders. These participants were randomized to receive assessments only in Stage 2, or were lost to follow up during Stage 1 and we not re-randomized during stage 2.
- MI-Only (Non-Responder): Participants randomized in Stage 1 two MI sessions focusing on stimulant use, sexual risk, and PrEP uptake delivered via Zoom. These participants were randomized to receive assessments only in Stage 2, or were lost to follow up during stage 1 and were not re-randomized during stage 2.
- CM+MI (Non-Responder): Sequential delivery of CM (Stage 1) and MI (Stage 2) for non-responders that were randomized in Stage 2 to "switch."
- MI+CM (Non-Responder): Sequential delivery of MI (Stage 1) and CM (Stage 2) for non-responders that were randomized in Stage 2 to "switch."
- CM-Only (Responder): Responders randomized to receive CM financial incentives for PrEP clinical evaluation and uptake in Stage 1 who provided evidence of a recent PrEP prescription.
- Total: Total of all reporting groups
Arm/Group | CM-Only (Non-Responder) | MI-Only (Non-Responder) | CM+MI (Non-Responder) | MI+CM (Non-Responder) | CM-Only (Responder) | MI-Only (Responder) | Total
Number analyzed (Participants) | 15 | 21 | 9 | 7 | 11 | 7 | 70
Age, Continuous [Geometric Mean (Standard Deviation); unit: Years] | 41 (9) | 41 (11) | 40 (8) | 45 (5) | 43 (10) | 36 (8) | 41 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 15 | 21 | 9 | 7 | 11 | 7 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 5 | 1 | 0 | 2 | 12
  Not Hispanic or Latino | 14 | 18 | 4 | 6 | 11 | 5 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 3 | 0 | 6
  White | 10 | 18 | 7 | 4 | 7 | 4 | 50
  More than one race | 3 | 0 | 1 | 1 | 1 | 1 | 7
  Unknown or Not Reported | 0 | 2 | 0 | 1 | 0 | 1 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 21 | 9 | 7 | 11 | 7 | 70
Annual Income [Count of Participants; unit: Participants] — Annual income in the past year
  Participants
    Less than $5,000 | 1 | 4 | 1 | 0 | 1 | 0 | 7
    $5,000 - $24,999 | 5 | 7 | 3 | 2 | 3 | 3 | 23
    $25,000 - $74,999 | 7 | 6 | 4 | 2 | 7 | 4 | 30
    $75,000 - $99,000 | 0 | 2 | 1 | 3 | 0 | 0 | 6
    $100,000 or more | 1 | 2 | 0 | 0 | 0 | 0 | 3
    Unknown | 1 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Filling a Prescription for PrEP
Description: The proportion of participants who provide evidence that they have filled a PrEP prescription
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Groups:
- CM-Only (Non-Responder or Lost to Follow Up During Stage 1): Participants randomized in Stage 1 to receive CM financial incentives for PrEP clinical evaluation and filling a PrEP prescription that were non-responders. These participants were randomized to receive assessments only in Stage 2, or were lost to follow up during Stage 1 and we not re-randomized during stage 2.
- MI-Only (Non-Responder or Lost to Follow Up During Stage 1): Participants randomized in Stage 1 two MI sessions focusing on stimulant use, sexual risk, and PrEP uptake delivered via Zoom.. These participants were randomized to receive assessments only in Stage 2, or were lost to follow up during stage 1 and were not re-randomized during stage 2.
- CM+MI: Sequential delivery of CM (Stage 1) and MI (Stage 2) for non-responders that were randomized in Stage 2 to "switch."
- MI+CM: Sequential delivery of MI (Stage 1) and CM (Stage 2) for non-responders that were randomized in Stage 2 to "switch."
- CM-Only (Responder): Randomized in Stage 1 to CM financial incentives for PrEP clinical evaluation and filling a PrEP prescription and provided evidence of a recent PrEP prescription.
- MI-Only (Responder): Randomized in Stage 1 to two MI sessions focusing on stimulant use, sexual risk, and PrEP use, and provided evidence of a recent PrEP prescription.
Arm/Group | CM-Only (Non-Responder or Lost to Follow Up During Stage 1) | MI-Only (Non-Responder or Lost to Follow Up During Stage 1) | CM+MI | MI+CM | CM-Only (Responder) | MI-Only (Responder)
Number analyzed (Participants) | 5 | 13 | 9 | 7 | 11 | 7
Participants
  Yes | 0 | 2 | 2 | 5 | 11 | 7
  No | 5 | 11 | 7 | 2 | 0 | 0

2. Secondary Outcome: Proportion of Participants Who Self-report PrEP Clinical Evaluation by a Medical Provider
Description: The proportion of participants reporting that they attended a medical appointment to be evaluated for PrEP.
Time Frame: 6 Months
Measure: Count of Participants; unit: Participants
Groups:
- Contingency Management (CM) - Only (Non-Responder): Participants randomized in Stage 1 to receive CM financial incentives for PrEP clinical evaluation and filling a PrEP prescription that were non-responders. These participants were randomized to receive assessments only in Stage 2.
- Motivational Interviewing (MI) - Only (Non-Responder): Participants randomized in Stage 1 two MI sessions focusing on stimulant use, sexual risk, and PrEP uptake delivered via Zoom.. These participants were randomized to receive assessments only in Stage 2.
Arm/Group | Contingency Management (CM) - Only (Non-Responder) | Motivational Interviewing (MI) - Only (Non-Responder) | CM+MI | MI+CM | CM-Only (Responder) | MI-Only (Responder)
Number analyzed (Participants) | 5 | 13 | 9 | 7 | 11 | 7
Participants
  Yes | 3 | 9 | 8 | 4 | 11 | 7
  No | 2 | 4 | 1 | 3 | 0 | 0

3. Secondary Outcome: Clinical Cut Points for Self-reported Methamphetamine Use Severity
Description: Participants will complete the Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST), which provides validated composite scores indexing the severity of methamphetamine use (Mild = 0-3; Moderate = 4-26; Severe = 27 or greater).
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Contingency Management (CM) - Only (Non-Responder) | Motivational Interviewing (MI) - Only (Non-Responder) | CM+MI | MI+CM | CM-Only (Responder) | MI-Only (Responder)
Number analyzed (Participants) | 3 | 12 | 8 | 5 | 7 | 7
Participants
  Mild (0-3) | 2 | 7 | 2 | 4 | 2 | 6
  Moderate (4-26) | 1 | 1 | 6 | 0 | 3 | 0
  Severe (27 or greater) | 0 | 4 | 0 | 1 | 2 | 1

4. Secondary Outcome: Proportion of Participants Who Reported Receptive Condomless Anal Sex (Receptive CAS)
Description: Participants will complete a detailed behavioral assessment to report the number of men with whom they have had receptive CAS. The proportion of participants reporting any receptive CAS will be reported.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Contingency Management (CM) - Only (Non-Responder) | Motivational Interviewing (MI) - Only (Non-Responder) | CM+MI | MI+CM | CM-Only (Responder) | MI-Only (Responder)
Number analyzed (Participants) | 3 | 12 | 8 | 5 | 7 | 7
Participants
  Yes | 0 | 6 | 4 | 2 | 2 | 3
  No | 3 | 6 | 4 | 3 | 5 | 4

5. Secondary Outcome: Proportion of Participants Who Reported Insertive Condomless Anal Sex (Insertive CAS)
Description: Participants will complete a detailed behavioral assessment to report the number of men with whom they have had insertive CAS. The proportion of participants reporting any insertive CAS will be reported.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Contingency Management (CM) - Only (Non-Responder) | Motivational Interviewing (MI) - Only (Non-Responder) | CM+MI | MI+CM | CM-Only (Responder) | MI-Only (Responder)
Number analyzed (Participants) | 3 | 12 | 8 | 5 | 7 | 7
Participants
  Yes | 2 | 6 | 4 | 2 | 5 | 6
  No | 1 | 6 | 4 | 3 | 2 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each participant for 6 months.
Description: The AEs and SAEs conformed to standard definitions for clinicaltrials.gov.
Groups:
- CM - Non-Responder: Contingency Management (CM): CM will include financial incentives for PrEP clinical evaluation and filling a PrEP prescription.
- MI - Non-Resonder: Motivational Interviewing (MI): Two MI counseling sessions focusing on stimulant use, sexual risk, and PrEP uptake will be delivered via Zoom.
- CM+MI: Sequentially delivered CM+MI for non-responders who were randomized at the stage-two randomization to switch to the other condition.
- MI+CM: Sequentially delivered MI+CM for non-responders who were randomized at the stage-two randomization to switch to the other condition.
- CM - Responder: Contingency Management (CM): CM will include financial incentives for PrEP clinical evaluation and filling a PrEP prescription. These participants responded before Stage 2 randomization.
- MI - Responder: Motivational Interviewing (MI): Two MI counseling sessions focusing on stimulant use, sexual risk, and PrEP uptake will be delivered via Zoom. These participants responded before Stage 2 randomization.
Arm/Group | CM - Non-Responder | MI - Non-Resonder | CM+MI | MI+CM | CM - Responder | MI - Responder
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/21 | 0/9 | 0/7 | 0/11 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/21 | 0/9 | 0/7 | 0/11 | 0/7
Other Adverse Events (participants affected / at risk) | 0/15 | 0/21 | 0/9 | 0/7 | 0/11 | 0/7

LIMITATIONS AND CAVEATS:
This was a pilot sequential multiple assignment randomized trial (SMART) of sequentially delivered CM and MI interventions. Only non-responders after three months (i.e., those who had not started or restarted PrEP) were randomized to Switch or Continue with assessments only. Given the sample size and sequential randomization, effect sizes should be interpreted with caution. In fact, the most appropriate purpose of a pilot trial is feasibility and acceptability to guide a more definitive trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT04205487/Prot_ICF_001.pdf
  • Statistical Analysis Plan (2024-08-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT04205487/SAP_002.pdf